CLINICAL TRIAL: NCT06783153
Title: Efficacy and Safety of Adjunctive Use of Rifaximin In Preventing Radiotherapy-induced Diarrhea in Cancer Patients
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Noha Mansour, Associate professsor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-238
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Radiotherapy Induced Diarrhea; Acute Radiation Enteritis; Prostate Cancer; Cervical Adenocarcinoma; Bladder (Urothelial, Transitional Cell) Cancer; Rectal Adenocarcinoma; Pelvic Radiotherapy; Rifaximin
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Rectal Neoplasms | interventions — Rifaximin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (Active Comparator)
  Interventions: Drug: Standard Care Chemoradiation
- Patients will receive Rifaximin 550 MG in addition to Pelvic Radiotherapy with/not chemotherapy (Experimental)
  Interventions: Drug: Rifaximin 550 MG

INTERVENTIONS:
Drug: Rifaximin 550 MG — Oral Rifaximin 550mg twice daily from the start of pelvic radiotherapy, with or without chemotherapy, as a preventive measure, and continuing every day until the end of the treatment up to 5 to seven weeks.
  Arms: Patients will receive Rifaximin 550 MG in addition to Pelvic Radiotherapy with/not chemotherapy
Drug: Standard Care Chemoradiation — Patients will receive standard chemotherapy and/or radiation
  Arms: Control Arm

SUMMARY:
Preclinical data indicate that rifaximin could be repurposed as a novel strategy for preventing and reducing the severity of gastrointestinal damage, particularly diarrhea, that results from pelvic irradiation. So, The aim of the work is to investigate the impact of Rifaximin on the incidence and severity of radiotherapy-induced diarrhea in cancer patients undergoing pelvic irradiation with or without chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are 18 years of age or older and have been diagnosed with non metastatic pelvic cancers.
* Patients who are undergoing curative intent radiotherapy with or without chemotherapy treatment.

Exclusion Criteria:

* Patients who have a record of intestinal resection in their medical history.
* Patients with a medical background of irritable bowel syndrome.
* Patients with a history of inflammatory bowel disease.
* Patients who regularly take anti-diarrheal medications before commencing radiotherapy.
* Patients experiencing diarrhea at the outset of the study.
* Patients with compromised immune systems, such as those who are HIV positive or using immunosuppressive medications.
* Pregnant or lactating woman.
* Patients allergic to rifamycin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The difference in the incidence and severity of radiotherapy induced diarrhea grade 2 or more according to Common Terminology Criteria for Adverse Events (CTCAE)in cancer patients undergo pelvic irradiation. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Province, Egypt